CLINICAL TRIAL: NCT01775358
Title: A Randomized, Single-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety and Tolerability of ALRN-5281 Administered by Subcutaneous Injection in Healthy Adult Volunteers
Brief Title: Phase 1 Safety Study of ALRN-5281 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aileron Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ALRN-100-01
Record Dates: First submitted 2013-01-17; First posted 2013-01-25 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- ALRN-5281 0.015 mg/kg (Experimental): Dosage-0.015 mg/kg
  Interventions: Drug: ALRN-5281 0.015 mg/kg
- ALRN-5281 0.05 mg/kg (Experimental): Dosage- 0.05 mg/kg
  Interventions: Drug: ALRN-5281 0.05 mg/kg
- ALRN-5281 0.15 mg/kg (Experimental): Dosage- 0.15 mg/kg
  Interventions: Drug: ALRN-5281 0.15 mg/kg
- Placebo 0.015 mg/kg (Placebo Comparator): Dosage- 0.015 mg/kg
  Interventions: Drug: Placebo 0.015 mg/kg
- Placebo 0.05 mg/kg (Placebo Comparator): Dosage- 0.05 mg/kg
  Interventions: Drug: Placebo 0.05mg/kg
- Placebo 0.15 mg/kg (Placebo Comparator): Dosage - 0.15 mg/kg
  Interventions: Drug: Placebo 0.15mg/kg

INTERVENTIONS:
Drug: ALRN-5281 0.015 mg/kg
  Arms: ALRN-5281 0.015 mg/kg
Drug: ALRN-5281 0.05 mg/kg
  Arms: ALRN-5281 0.05 mg/kg
Drug: ALRN-5281 0.15 mg/kg
  Arms: ALRN-5281 0.15 mg/kg
Drug: Placebo 0.015 mg/kg
  Arms: Placebo 0.015 mg/kg
Drug: Placebo 0.05mg/kg
  Arms: Placebo 0.05 mg/kg
Drug: Placebo 0.15mg/kg
  Arms: Placebo 0.15 mg/kg

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of a single dose of ALRN-5281 administered by subcutaneous injection to healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects aged 20 to 50 years, inclusive, at the time of informed consent.
2. Subjects must be in good health as determined by the Investigator based on detailed medical history, physical examination, vital signs, clinical laboratory tests, ECGs and other screening evaluations.
3. Ability to provide written informed consent and complying with all study requirements and restrictions.
4. Is a non-smoker and non-tobacco user for a minimum of 6 months prior to screening

Exclusion Criteria:

1. History or current evidence of any clinically significant cardiac, endocrinologic, hematologic, hepatobiliary, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, or other major disease, as determined by the Investigator
2. Previous treatment with any GH Releasing Hormone (GHRH) analog.
3. Participation in another clinical trial or treatment with an investigational agent within 30 days or 5 half-lives, whichever is longer, prior to enrollment.
4. History of cancer within the past five years (excluding non-melanoma skin cancer).
5. History of alcohol or drug abuse or dependence within 12 months of screening as determined by the Investigator.
6. Subjects with a body weight > 120 kg.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 28 days

SECONDARY OUTCOMES:
Serum IGF-1 | Predose, Day 1-Day 28
Serum GH | Predose, Day 1-Day 28
Time to Reach Maximum Observed Plasma Concentration (Tmax) of ALRN-5281 | Predose, Day 1- 0.5,1,2,3,4,6,8,10,12,14 and 16hr post dose , Day 2-Day11 and Day14
Maximum plasma concentration (Cmax) of ALRN-5281 | Predose, Day 1- 0.5,1,2,3,4,6,8,10,12,14 and 16hr post dose , Day 2-Day11 and Day14
Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] | Pre Dose, Day1- 0.5,1,2,3,4,6,8,10,12,14 and 16h post dose, Day2- Day11 and Day 14
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley D Vince, D.O., Principal Investigator — Vince and Associates; Hubert C Chen, M.D., Study Director — Aileron Therapeutics, Inc.
Locations (1):
- Vince and Associates Clinical Research, LLC, Overland Park, Kansas, United States